CLINICAL TRIAL: NCT03082950
Title: Influence of Hpv Infections on Therapeutical Outcome of Patients Suffering From Vulvar Cancer and Ist Preinvasive Lesions
Brief Title: HPV Infections, Cancer of the Vulva and Therapeutical Success
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Collaborators: EUROIMMUN Medizinische Labordiagnostika AG (Unknown)
Responsible Party: Principal Investigator, Daniel Alexander Beyer, University of Luebeck, University of Luebeck
Other Study IDs: HL-15-220
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: HPV; Human Papilloma Virus
Keywords: hpv prevalence; recurrence rate; survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tumor tissue samples are analyzed according to their hpv status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: human papilloma Virus (hpv) associated vulvar cancer incl. preinvasive lesions
  Interventions: Diagnostic Test: polymerase chain reaction
- 2: non-human papilloma Virus (hpv) associated vulvar cancer incl. preinvasive lesions
  Interventions: Diagnostic Test: polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: polymerase chain reaction — PCR is performed with all patients. The result (hpv positive or negative) will define the patiens Group Affiliation.
  Other Names: EUROARRAY

SUMMARY:
HPV infections may be responsible for different types of cancer in females. Primary Goal of the study was to identify the prevalence of an hpv affiliation in retrospective-prospective analysed cohort of patients who suffer from vulvar cancer and their preinvasive lesions.

DETAILED DESCRIPTION:
HPV infections may be responsible for different types of cancer in females. Primary Goal of the study was to identify the prevalence of an hpv affiliation in retrospective-prospective analysed cohort of patients who suffer from vulvar cancer and their preinvasive lesions.

After having retrospectively identified patients with vulvar cancer incl. their preinvasive lesions in the clinical registry the hpv status of the samples is prospectively analyzed using a new multiplex pcr Array. Two Groups are build: patients with hpv associated vulvar cancer and patients with non-hpv associated vulvar cancer.

Then, the rate of patients who respond to radiotherapy within the Groups is analyzed by building Kaplan meier plots according to the patients survival and recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* pts. who suffer from vulvar cancer and their preinvasive lesions
* positive informed consent
* complete set of data
* Treatment in luebeck university

Exclusion Criteria:

* opposite of above

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female the illness only affiliates females
Study Population: pts. who suffer from vulvar cancer and their preinvasive lesions who were treated in luebeck University medical Center over a 15 year period
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
prevalence of hpv infections among pations suffering from vulvar cancer and preinvasive lesions | 15yrs

SECONDARY OUTCOMES:
disease free survival among the groups | 15yrs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Beyer, MD, Principal Investigator — Westpfalz-Klinikum
Locations (1):
- Luebeck University, Department for obstetrics and gynecology, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Massad LS, Jeronimo J, Katki HA, Schiffman M; National Institutes of Health/American Society for Colposcopy and Cervical Pathology Research Group. The accuracy of colposcopic grading for detection of high-grade cervical intraepithelial neoplasia. J Low Genit Tract Dis. 2009 Jul;13(3):137-44. doi: 10.1097/LGT.0b013e31819308d4. PMID 19550210
- [Background] Sri T, Merideth MA, Pulanic TK, Childs R, Stratton P. Human papillomavirus reactivation following treatment of genital graft-versus-host disease. Transpl Infect Dis. 2013 Aug;15(4):E148-51. doi: 10.1111/tid.12098. Epub 2013 May 28. PMID 23710698
- [Background] Nocon M, Mittendorf T, Roll S, Greiner W, Willich SN, von der Schulenburg JM. Review on the medical and health economic evidence for an inclusion of colposcopy in primary screening programs for cervical cancer. GMS Health Technol Assess. 2007 Aug 10;3:Doc07. PMID 21289941